CLINICAL TRIAL: NCT06124066
Title: THE EFFECTS OF MIRABEGRON AND TAMSULOSIN FOR PATIENTS WITH URETERAL STENTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Muhammad Asykar Palinrungi, Head of Division of Urology, Department of Surgery, Faculty of Medicine, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 583/UN4.6.4.5.37/PP36/2022
Record Dates: First submitted 2023-09-02; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ureteral Stone; Kidney Stones; Ureteral Stenosis
Keywords: Double J stent; Mirabegron; Tamsulosin; Interleukin-6; Interleukin-10; lower urinary tract symptoms
MeSH Terms: conditions — Ureterolithiasis; Kidney Calculi; Lower Urinary Tract Symptoms | interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 3 groups of drug administration: Group A, Group B, and Group C.
Who Masked: Investigator
Masking Description: All medicines were placed in the same 3 boxes, which were held by the paramedics so that the patients and paramedics did not know the allocation of the types of drugs given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirabegron (Active Comparator): The participants were given mirabegron 50 mirabegron/day started 3 days before DJ stent insertion and until 6 weeks after the DJ stent insertion and filled in USSQ every week until 6 weeks after the DJ stent insertion(filled in directly when the patient arrived or by telephone)
  Interventions: Drug: Mirabegron 50 MG
- Tamsulosin (Active Comparator): The participants were given tamsulosin 0.4 mg that was started 3 days before DJ stent insertion and until 6 weeks after the DJ stent insertion and filled in USSQ every week until 6 weeks after the DJ stent insertion(filled in directly when the patient arrived or by telephone)
  Interventions: Drug: Mirabegron 50 MG
- Placebo (Placebo Comparator): The participants were given a placebo that was started 3 days before DJ stent insertion and until 6 weeks after the DJ stent insertion and filled in USSQ every week until 6 weeks after the DJ stent insertion(filled in directly when the patient arrives or by telephone)
  Interventions: Drug: Mirabegron 50 MG

INTERVENTIONS:
Drug: Mirabegron 50 MG — The participants were given mirabegron 50 mg or tamsulosin 0.4 mg and filled in the Ureteral Stent Symptom Questionnaire (USSQ), filled in directly when the patient arrived or by telephone.
  Other Names: Tamsulosin 0.4 mg; Placebo

SUMMARY:
Double J stent (ureteral stent) can cause discomfort to patients, generally due to irritation of the bladder mucosa, especially in the trigone area, smooth muscle spasm, and reflux of urine into the ureter. Complaints often appear in patients, especially lower urinary tract symptoms (LUTS), pain in the waist when urinating due to reflux of urine, sexual dysfunction, and hematuria.

Currently, to assess complaints after ureteral stent placement, the Ureteral Stent Symptom Questionnaire instrument consists of 6 topics: urinary complaints, pain, general health, work, sexual problems, and other things.

Interleukin-6 is an important inflammatory cytokine when irritation occurs after ureteral stent placement. Interleukin 10 is a cytokine with potent anti-inflammatory properties that plays a central role in limiting the host's immune response to pathogens, thereby preventing host damage and maintaining normal tissue homeostasis. The profile of these biomarkers has the potential to determine the correct prognosis and therapy.

Mirabegron is a β3 adrenergic receptor agonist that has a dual antioxidant effect that plays a key role in the first step of the antimicrobial response and early resolution of inflammation so that post-stent complaints similar to overactive bladder complaints can be resolved. Tamsulosin (a selective α1A- and α1D-adrenoceptor antagonist) has a relaxing effect on the smooth muscle in the prostate, the neck of the bladder, and the distal ureter, thereby reducing the inflammatory reaction and improving oxidative stress by reducing the formation of reactive oxidative stress.

DETAILED DESCRIPTION:
The research design used was experimental with randomized sampling, double-blinded, in men and women with ureteral stents. The patient signed informed consent regarding blood and urine sampling, bladder mucosal biopsy, placement and removal of ureteral stents, drug administration, and side effects of therapy. The history and physical examination of the patient were recorded including age, height, weight, and body mass index (BMI). Investigation procedures for urinalysis, routine blood, SGOT/SGPT, urea/creatinine, blood sugar during, ultrasonography, plain abdominal photos, and CT scan urography were performed on patients before surgery. The patient's largest stone size is used as a benchmark to record the patient's stone size.

All patients who underwent routine post-ureterorenoscopy lithotripsy (URSL) ureteral stent procedures and met the inclusion and exclusion criteria were included in the study evaluation. The ureteral stent used was 4.7 Fr in size with a length of 24-26 cm, made from polyurethane used in all patients.

Blood and urine samples will be taken before drug administration begins, and when the ureteral stent is removed or replaced. Bladder mucosal biopsy was performed in the trigone vesicae around the contralateral ureteral opening during cystoscopy before ureteral stent placement, and on the ipsilateral side when the ureteral stent was to be removed or replaced in the 6th week after ureteral stent placement.

A plain photo of the abdomen or ultrasound is done postoperatively to see the remaining stone fragments and the position of the ureteral stent. Urethral catheters were removed on the 2nd postoperative day in all patients before the patients were discharged and given oral antibiotics (cefadroxil) for 5 days. During the observation phase, the patient was given the same analgesic (paracetamol 500 mg every 8 hours/24 hours and if needed can be given every 6 hours/24 hours). The total amount of analgesics consumed by the patient will be recorded in filling out the final questionnaire.

Patients were asked to come to the urology clinic at the hospital for control on the seventh day. The patient will be given a questionnaire format that will measure the presence or absence and severity of side effects experienced by the patient for 7 days after ureteral stent placement.

Patients will be divided into 3 groups of drug administration. The double-blinded method is used to minimize bias. All medicines were placed in the same 3 boxes, which were held by the paramedics so that the patients and researchers did not know the allocation of the types of drugs given. All patients have been informed about the side effects of the drug.

Administration of mirabegron 50 mg/day compared to tamsulosin 0.4 mg and placebo began on the third day before insertion of the ureteral stent. Completion of the questionnaire began on the seventh day after ureteral stent insertion, then it was measured every 7 days (7th, 14th, 21st, 28th, 35th, and 42nd day) after ureteral stent insertion. Filling out the questionnaire can be done by in-person interview at the clinic or by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient with first ureterorenoscopy and ureteral stent placement
* Using a semi-rigid (rigid) retrograde or flexible (flexible) ureteroscope
* Stent placement on one side
* Stent installation size 4.7 Fr, length 24-26cm hydrophilic coated ureteric stent
* Patients who can read and understand Indonesia language (Bahasa Indonesia)

Exclusion Criteria:

* Patients with or who have a history of malignancy of the urinary tract
* Patients with LUTS caused by benign prostatic enlargement, bladder stones, or urethral strictures
* Catheterized patients or on self-catheter therapy regularly and patients with urinary diversion
* Patients with Post void residual volume > 350 mL
* Patients with neurogenic bladder and/or OAB syndrome, stress incontinence, or mixed stress/urge incontinence
* Patients with chronic pain that is not controlled or on therapy to manage chronic pain
* Patients with symptomatic UTI
* Patients with a prior history of sexual dysfunction
* Have or are currently undergoing radiation therapy/hormonal therapy and/or surgical procedures in the minor pelvis, ureteral reconstructive surgery.
* Patients with primary neurological disorders, such as multiple sclerosis, Parkinson's disease, diabetic nephropathy, or other neurological diseases that affect bladder function.
* Patients who are hypersensitive to mirabegron and tamsulosin or their derivatives and patients with mirabegron and tamsulosin contraindications.
* The patient could not follow the research protocol due to an organic brain disorder or psychiatric disorder
* Patients with autoimmune diseases and other inflammatory diseases, as well as patients taking immunosuppressant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
serum and urine Interleukin-6 serum level (ELISA) | Pre-intervention and immediately after the intervention
  Interleukin-6 serum level
serum and urine Interleukin-10 serum level (ELISA) | Pre-intervention and immediately after the intervention
  Interleukin-10 serum level
Histopathology | Pre-intervention and immediately after the intervention
  The severity of the mucosal inflammatory reaction was graded using a semiquantitative scale where 0=none, 1 = focal lymphocytic infiltration, 2 =diffuse predominantly lymphocytic infiltration, 3 =diffuse predominantly eosinophil polymorphonuclear infiltration and 4 = grade 3 changes in combination with intra-epithelial eosinophilic micro-abscesses.
Urinary symptoms in the Ureteral Stent Symptom Questionnaire (USSQ) parameter | Pre-intervention, immediately after the interventio, and up to 4 weeks
  Minimum values 2 and maximum values 47

SECONDARY OUTCOMES:
Basis data | pre-intervention
  Characteristic data participants

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Palinrungi, Study Director — Hasanuddin University Hospital
Locations (1):
- DR Wahidin Sudirohusodo Hospital, Hasanuddin University Hospital, and Akademis Jaury Jusuf Putra Hospital., Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
The data supporting this study's findings are available on request from the corresponding author (Muhammad Asykar Palinrung).